CLINICAL TRIAL: NCT06874426
Title: The Impact of Endoscopic Endonasal Skull Base Surgery on Olfaction
Acronym: Endo-Olfact
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Laura Van Gerven, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S69823
Record Dates: First submitted 2025-02-11; First posted 2025-03-13 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Meningioma; Pituitary Disease; Pituitary Adenoma; Craniopharyngioma; Endoscopic Pituitary Surgery; Olfactory Dysfunction
Keywords: olfactory dysfunction; trigeminal dysfunction; endoscopic endonasal skull base surgery; pituitary surgery
MeSH Terms: conditions — Meningioma; Pituitary Diseases; Pituitary Neoplasms; Craniopharyngioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mucosa of the posterior part of the septum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic endonasal skull base surgery — This intervention will be performed as part of the standard-of-care for patients scheduled for endoscopic endonasal skull base surgery for lesions in the (para)sellar region
  Other Names: endoscopic pituitary surgery; anterior skull base surgery

SUMMARY:
In this study, the research team will investigate the incidence and etiology of olfactory dysfunction following endoscopic endonasal skull base surgery, by combining clinical assessments with histomolecular analysis.

DETAILED DESCRIPTION:
The incidence of olfactory dysfunction following endoscopic endonasal skull base surgery remains unclear in current research, and the results vary widely. Additionally, the pathophysiology of this postoperative olfactory dysfunction and the impact of this surgery on the trigeminal system has not been investigated to date. In this study, the investigators developed a state-of-the-art clinical pipeline with olfactory and trigeminal assessments, prior to and following endoscopic endonasal skull base surgery. Furthermore, the investigators will collect surgical waste tissue from the posterior septal mucosa, which is removed during this procedure to gain access to the sphenoid sinus and the (para)sellar region. By performing histomolecular analysis, the research group aims to elucidate the pathophysiology of olfactory dysfunction following this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for endoscopic endonasal skull base surgery

Exclusion Criteria:

* Pre-existing anosmia
* Patients has a history of previous endoscopic endonasal skull base surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with an indication for endoscopic endonasal skull base surgery for lesions in the anterior skull base (the parasellar region)
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of olfactory dysfunction | From enrollment to the last evaluation 6 months postoperatively
Incidence of trigeminal dysfunction | From enrollment to the last evaluation 6 months postoperatively
Etiology of olfactory and trigeminal dysfunction following endoscopic endonasal skull base surgery | Until the end of study (at 3 years)

SECONDARY OUTCOMES:
Risk factors for olfactory dysfunction following endoscopic endonasal skull base surgery | From enrollment to the last evaluation 6 months postoperatively
  Parameters such as smoking history, allergies, age, gender, co-morbidities will be investigated as possible covariates

CONTACTS AND LOCATIONS:
Locations (3):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium
- Max Planck Research Unit for Neurogenetics, Frankfurt am Main, Hesse, Germany
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided